CLINICAL TRIAL: NCT03650101
Title: Improving Infant Hydrocephalus Outcomes in Uganda: Predicting Developmental Outcomes and Identifying Patients at Risk for Early Treatment Failure After ETV/CPC
Brief Title: Improving Infant Hydrocephalus Outcomes in Uganda
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); CURE Children's Hospital, Uganda (Other); Yale University (Other)
Responsible Party: Principal Investigator, Pei-Yi Lin, Assistant Professor, Boston Children's Hospital
Other Study IDs: P00029806
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hydrocephalus group: Inclusion criteria:
  1. Age less than six months
  2. Symptomatic hydrocephalus characterized by abnormal rate of head growth, full anterior fontanel, ventriculomegaly
  3. A parent or a guardian qualified by Ugandan law to give informed consent
  4. Patients from Eastern, Central and Northern districts of Uganda, and in geographic proximity to CURE hospital will be eligible
  Exclusion criteria:
  1. Age greater than six months
  2. No evidence of progressive hydrocephalus
  3. Patients outside of the districts specified in the inclusion criteria
  Interventions: Procedure: ETV/CPC
- Control group: Inclusion criteria:
  1. Born at GA ≥ 37 weeks
  2. Age less than six months at the time of enrollment
  3. No known medical conditions
  4. With a parent or a guardian qualified by Ugandan law to give informed consent
  5. Parents live in one of the villages in the Mbale or Budaka District, in geographic proximity to CCHU.
  Exclusion criteria:
  1. Born at GA < 37 weeks
  2. Age greater than six months
  3. Evidence of one or more medical conditions
  4. Living outside of the districts specified in the inclusion criteria.

INTERVENTIONS:
Procedure: ETV/CPC — The Endoscopic Third Ventriculostomy/Choroid Plexus Cauterization (ETV/CPC) will comprise a standard frontal approach with flexible endoscopy.
  Groups: Hydrocephalus group

SUMMARY:
Neonatal postinfectious hydrocephalus (PIH) is a major public health problem in East Africa.The standard treatment has long been placement of a ventriculoperitoneal shunt (VPS) but these devices require life-long maintenance and nearly all fail multiple times. Endoscopic Third Ventriculostomy (ETV) with Choroid Plexus Cauterization (ETV/CPC) is an alternate treatment to give patients a shunt-free life. In this study, the investigators aim to optimize the metrics of evaluation as quantitative prognostic indicators of treatment response and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 180 days (six months) old
* Symptomatic hydrocephalus characterized by abnormal rate of head growth, full anterior fontanel, ventriculomegaly
* A parent or a guardian qualified by Ugandan law to give informed consent
* Patients from Eastern, Central and Northern districts of Uganda, and in geographic proximity to CURE hospital will be eligible

Exclusion Criteria:

* Age greater than six months
* No evidence of progressive hydrocephalus
* Patients outside of the districts specified in the inclusion criteria

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants less than six months old with progressive hydrocephalus
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant Development, Third Edition (BSID-3), cognitive scaled score | 24 months of age
  Scores on the BSID-3, which is used to evaluate infants and toddlers 1 to 42 months of age, range from 1 to 19, with higher scores indicating better performance; the mean (±standard deviation(SD)) score in the general population is 10±3.
Incidence of ETV/CPC treatment failure | 6 months post-treatment
  Treatment failure or success will be determined with the use of clinical and radiographic criteria.
  * Treatment success will be determined as the shift in the growth of head circumference to a normal rate, as plotted on a standard growth chart; decompression of the anterior fontanel; relief of symptoms of elevated intracranial pressure, such as irritability and vomiting; resolution of down-gaze or sixth cranial nerve palsy; and a decrease or arrest in ventriculomegaly as determined on Computerized Tomography (CT).
  * Treatment failure will be defined as treatment-related death or the need for a second operation for infection or for the recurrence of hydrocephalus.

SECONDARY OUTCOMES:
Cerebral oxygen metabolism | pre- and post-, 6, 12 months post-treatment and 24 months of age
  cerebral oxygen metabolism will be measured with near-infrared spectroscopy
brain volume | pre-, 6, 12 months post-treatment and 24 months of age
  brain volume will be quantitatively estimated from the head CT scan
Bayley Scales of Infant Development, Third Edition (BSID-3), cognitive scaled score at 12 months post-treatment | 12 months post-treatment
  Scores on the BSID-3, which is used to evaluate infants and toddlers 1 to 42 months of age, range from 1 to 19, with higher scores indicating better performance; the mean (±standard deviation) score in the general population is 10±3.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yi Lin, PhD, Principal Investigator — Boston Children's Hospital
Locations (3):
- Penn State University, University Park, Pennsylvania, United States
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Cure Children's Hospital of Uganda, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside of the study team.

REFERENCES:
- [Result] Vadset TA, Rajaram A, Hsiao CH, Kemigisha Katungi M, Magombe J, Seruwu M, Kaaya Nsubuga B, Vyas R, Tatz J, Playter K, Nalule E, Natukwatsa D, Wabukoma M, Neri Perez LE, Mulondo R, Queally JT, Fenster A, Kulkarni AV, Schiff SJ, Grant PE, Mbabazi Kabachelor E, Warf BC, Sutin JDB, Lin PY. Improving Infant Hydrocephalus Outcomes in Uganda: A Longitudinal Prospective Study Protocol for Predicting Developmental Outcomes and Identifying Patients at Risk for Early Treatment Failure after ETV/CPC. Metabolites. 2022 Jan 14;12(1):78. doi: 10.3390/metabo12010078. PMID 35050201